CLINICAL TRIAL: NCT06152211
Title: Using Music-Based Interventions to Improve the Quality of Life and Wellbeing of Older Adults With or at Risk of Alzheimer's Disease
Brief Title: Music-Based Interventions, Aging, Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Assal Habibi, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APP-23-05720
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Speech Perception; Anxiety; Social Behavior
Keywords: music, choir, aging, dementia, APOE ε4
MeSH Terms: conditions — Anxiety Disorders; Social Behavior; Dementia

STUDY DESIGN:
Intervention Model Description: An individually randomized group treatment trial where adults ages 65 and older half of carriers of APOE ε4 and the other half of non-carriers will be randomly assigned to a 16-week: (1) community choir program or (2) a group music listening program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be masked to the hypothesis of the study. Outcome assessors and investigators will be masked to the group randomization. Randomization will be stratified on gender, age (<77, ≥77), APOE ε4 carrier status, and hearing aid use. The randomization list will be prepared by an expert statistician outside of the study team.One one research coordinator will have access to the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choir (Experimental): For each choir session, the choir director will be supported by an accompanist who will provide the music accompaniment for the songs and four section leaders who will provide musical leadership for choral sections (soprano, alto tenor & bass). At the beginning of each choir group, participants will be asked about their favorite songs to help ensure that the music will be appropriate for the participants' interest and cultural background. Each choir group will rehearse once a week for two hours with a short break in the middle for snacks for a total of 16 consecutive weeks. The choir rehearsals will follow a general routine, beginning with announcements and warm-ups, work on the repertoire, a break, additional work on the repertoire in sections, and a short group practice at the end. Participants will also be given at-home activities, in the form of pre-recorded videos and music theory exercises to complete outside of class for an estimated 1.5 hours per week.
  Interventions: Behavioral: Choir
- Music Listening (Active Comparator): Over the course of 16-weeks, the group will meet for two hours per week to talk about a set of musical recordings. Recorded music will be previously assigned and provided as a playlist via a web platform to track the time duration of engagement. Regular attendance will be required. The discussion group will meet as a full group each week to listen to a subset of that week's recordings, with a guided and brief discussion after each of the six selected songs. The group will then pause for a brief break and will divide into four smaller discussion groups where a volunteer facilitator from that group would guide a discussion about the selected music, to include personal reflections, its cultural context, and ideas around societal impacts.
  Interventions: Behavioral: Group Music Listening

INTERVENTIONS:
Behavioral: Choir — A choir for older adults is a musical/singing ensemble composed of individuals aged 65 and above. The choir rehearsals are weekly, 2 hours each and the length of the intervention is 16 weeks total.
  Other Names: Group Singing
  Arms: Choir
Behavioral: Group Music Listening — A weekly collective music listening, 2 hours each for 16 weeks.
  Arms: Music Listening

SUMMARY:
Using a randomized controlled trial design, the investigators will examine the effects of music engagement through choir training on the hearing, communication, and psychosocial well-being of older adults, particularly those at heightened risk of developing dementia.

DETAILED DESCRIPTION:
Major demographic transitions are underway in the developed world and adults aged 65 and over are the fastest growing segment of the United States population. Aging is associated with the deterioration of sensory and perceptual processes as well as a decline in cognitive functioning including attention and working memory. Advancing age is also associated with an increased risk of developing dementia including Alzheimer's disease (AD), a progressive neurodegenerative condition. The ε4 allele of APOE is one of three common alleles generated by cysteine/arginine substitutions. Although multiple genetic and environmental risk factors are involved in AD, the possession of the ɛ4 allele is recognized as the most common identifiable genetic risk factor for late-onset AD. The proportion of patients with AD that is attributable to the APOE ε4 is estimated to be 20% in people aged ≥ 55 years 5. Although the APOE 4 allele increases the risk of developing AD by three to fifteen times, recent studies have shown that the risk can be modified by non-genetic factors, including high education and leisure activities.

Another significant and related problem of aging is a decline in hearing abilities. Age-related hearing loss is a common problem for older adults, leading to communication difficulties, isolation, and cognitive decline. The difficulty understanding speech in noisy environments is one consequence of hearing loss that is particularly difficult to restore with hearing aids. Speech-in-noise (SIN) perception appears to be supported by both the efficiency of bottom-up sound encoding and the influence of higher-level top-down processes such as auditory working memory and selective attention. Decline in hearing and reduction in communication are associated with an increased rate of cognitive decline and the development of dementia in older adults. Decline in SIN perception can also make it difficult for aging individuals to engage socially and maintain relationships and has been linked to loneliness and depression. Indeed, poor SIN perception may contribute to cognitive decline and increased risk of dementia both through taxing cognitive load and decreasing social engagement. As a result, there is a critical need for effective and accessible interventions that target hearing, particularly interventions that are motivating and engaging and can be applied to the expanding population of older adults, especially those at higher risk of AD. The investigators will conduct an individually randomized group treatment trial to investigate the effects of choir training and its underlying neurobiological mechanisms on SIN perception and psychosocial well-being in adults ages 65 and older half carriers of APOE ε4 and the other half of non-carriers. The investigators will randomly assign approximately 66 older adults to a 16-week: (1) community choir program or (2) a group music listening program.

ELIGIBILITY:
Inclusion Criteria:

* Visual and Auditory Acuity: Adequate visual and auditory acuity, with correction if necessary.
* Language Proficiency: Fluency in English to ensure complete testing.

Exclusion Criteria:

* Hearing Loss: Severe hearing loss not correctable with aids.
* Neurological and Otologic Conditions: History of known neurological or otologic conditions.
* Psychiatric Disorders: Current severe psychiatric disorders (past disorders not included).
* Medical Conditions: Unstable or serious medical conditions that could limit participation in assessments or weekly meetings.
* Cognitive Function: Impaired cognitive function, indicated by a score of less than 26 on the Montreal Cognitive Assessment (MoCA).
* Music Training: Current or past professional music training, defined as 3 years of regular, formal practice, excluding typical educational curriculum music classes or singing in worship services.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Speech in Noise Perception ( SIN) as measured by QuickSIN | 16 weeks
  The ability to understand speech in noisy environments

SECONDARY OUTCOMES:
Self-Efficacy as measured by NIH Toolbox Self-Efficacy Short Form | 16 weeks
  Belief in one's capacity to have control over life events
Interest in Life as measured by Apathy Short Form measure from NIH Toolbox | 16 weeks
  Interest and engagement in life
Loneliness as measured by NIH Toolbox Loneliness Short Form | 16 weeks
  The degree to which a person is socially isolated from others

OTHER OUTCOMES:
Anxiety as measured by State Trait Anxiety Inventory for Adults | 16 weeks
  anxiety symptoms
Auditory Encoding as measured by auditory evoked potentials N1, P2 and P3 (EEG) | 16 weeks
  Strength of encoding auditory stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All study protocols and analysis plans will be shared. Raw EEG data will be made available in its original format that can be accessed and imported to different analysis software. A supplement document with additional information about protocol design and relevant triggers and responses will also be provided in the data dictionary.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following the NIH Data Sharing Policy and Implementation Guidelines, we plan to make the datasets available for sharing at the time that the main project findings are accepted for publication. That is, the raw data files and analysis scripts, which will initially be used for internal study team purposes, will be available for public use after our main intervention effects paper is published; within one year of the final year of funding.
Access Criteria: Individual researchers can contact the PIs for data and through filling out a data request and use form that we will create for the purposes of data sharing